CLINICAL TRIAL: NCT02850679
Title: Finnish Elective Cardioversion for Persistent Atrial Fibrillation Study
Brief Title: FINnish CardioVersion Study II
Acronym: FinCV2
Status: Completed | Type: Observational
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Juhani Airaksinen, Professor of Cardiology, University of Turku
Other Study IDs: T118/2014
Record Dates: First submitted 2016-07-26; First posted 2016-08-01 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Cardioversion
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a retrospective multi-center patient cohort study investigating patients with persistent atrial fibrillation (AF) and elective cardioversion (ECV). The aim is to identify clinical predictors for ineffective ECV to improve management quality of persistent AF.

DETAILED DESCRIPTION:
Data was gathered from patient registries of two finnish university hospitals and two regional hospitals in a time period of 2003-2015. A data search was conducted using the ICD-10 code for atrial fibrillation and NCSP code for cardioversion. All patients with AF and performed cardioversion were eligible for the study.

Initially, 2373 patients were captured after which all ECV cases were identified and included manually in the study using a structured electronic case report form. The study cohort comprised 1998 ECVs and 1342 patients. Follow-up data was gathered for 30 days after ECV and all strokes, transient ischemic attacks, arrhythmic complications, AF recurrences and failed cardioversions were recorded and subjected to careful exploration. IBM SPSS Statistics software version 22.0 was used to perform all analyses.

ELIGIBILITY:
Inclusion Criteria:

* All patients with persistent (>48h) atrial fibrillation and elective electrical cardioversion

Exclusion Criteria:

* Cardioversions for patients with acute (<48h) atrial fibrillation
* Pharmacological cardioversions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1342 patients with 1998 elective cardioversions
Sampling Method: Non-Probability Sample
Enrollment: 1342 (Actual)
Dates: Start 2014-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Fatal or Non-fatal Stroke/TIA | 30 days

SECONDARY OUTCOMES:
Arrhythmic Complications | 24 hours
  bradyarrhythmias, ventricular tachycardia and ventricular fibrillation
Failure of Cardioversion | 24 hours
  Assessed at discharge
Recurrence of AF after ECV | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Juhani Airaksinen, Professor, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: Undecided